CLINICAL TRIAL: NCT07120490
Title: Multicenter, Randomized, Open-label, Three-arm Study on the Efficacy of Fecal Microbiota Transplantation vs Fidaxomicin vs Vancomycin in the Treatment and Relapse Prophylaxis of Clostridioides Difficile Infection. STOP-CDI Study
Brief Title: STOP-CDI: Efficacy of Fecal Microbiota Transplantation vs Fidaxomicin vs Vancomycin in Treating and Preventing Relapse of Clostridioides Difficile Infection
Acronym: STOP-CDI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Human Biome S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP-CDI; 2022/ABM/03/00047 (Other Grant/Funding Number: Medical Research Agency)
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-03

CONDITIONS: Clostridioides Difficile Infection; Clostridioides Difficile Infection Recurrence; Fecal Microbiota Transplantation (FMT); Comparative Effectiveness of CDI Treatments; Fidaxomicin; Vancomycin
Keywords: Clostridioides difficile; CDI; Fecal microbiota transplantation; Fidaxomicin; Vancomycin; Recurrent infection
MeSH Terms: conditions — Clostridium Infections; Reinfection | interventions — Fecal Microbiota Transplantation; Fidaxomicin; Vancomycin; Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, open-label, three-arm study using a parallel assignment model. Eligible participants are randomly allocated in a 2:1:1 ratio to one of three intervention groups: (1) short-course oral vancomycin followed by fecal microbiota transplantation (FMT), (2) fidaxomicin monotherapy, or (3) standard-of-care vancomycin. Each participant remains in their assigned group for the duration of the study and receives only the intervention corresponding to that group. No crossover between arms is planned. The parallel design allows for direct comparison of recurrence rates and treatment outcomes across independent, concurrently treated cohorts. Randomization is stratified by site, and outcome assessors may be blinded for certain exploratory analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FECAL MICROBIOTA TRANSPLANTATION (with vancomycin short pretreatment phase) (Experimental): Participants receive oral vancomycin (125 mg QID) for 5 days (extendable to 10 if needed), followed by FMT. On Day 6, bowel cleansing is performed (macrogol-based), and biological samples (stool, blood, urine, saliva) are collected. On Day 7, FMT is administered via preferred oral capsules or, if necessary, colonoscopy, gastroscopy, NJ tube, or rectal enema. A second FMT is given either as daily capsules on Days 9-14 or as a single dose via other routes on Day 14. Dosing: 6 jars of capsules or 200 mL suspension (≥35 kg); half for <35 kg. Supportive measures include antiemetics and fasting. Oral non-antibiotic medications continue. Post-FMT samples are collected for follow-up analyses.
  Interventions: Other: FMT (fecal microbiota transplantation)
- ANTIBIOTICS ONLY - FIDAXOMICIN (Experimental): Participants receive fidaxomicin 200 mg twice daily for 10 days. Biological samples (stool, blood, urine, saliva) are collected at baseline (before first antibiotic dose) for microbiome and safety analyses (PRE ATB). No additional interventions are applied. The antibiotic eradication phase ends on Day 10, after which the participant enters the follow-up phase. Post-treatment biological samples are collected (POST ATB) to assess treatment response, recurrence risk, and microbiota changes.
  Interventions: Drug: Fidaxomicin
- ANTIBIOTICS ONLY - VANCOMYCIN (Experimental): Participants receive vancomycin 125 mg four times daily for 10 days. Biological samples (stool, blood, urine, saliva) are collected prior to the first dose (PRE ATB) for safety and exploratory analyses. No additional therapies are administered. The eradication procedure is completed on Day 10, followed by a post-treatment sampling phase (POST ATB) for assessment of recurrence, clinical response, and microbiome status.
  Interventions: Drug: Vancomycin (VAN) treatment

INTERVENTIONS:
Other: FMT (fecal microbiota transplantation) — This intervention consists of a two-phase treatment for Clostridioides difficile infection in high-risk adults. First, participants receive a short-course (5 days) of oral vancomycin to reduce C. difficile bacterial load. Following antibiotic pretreatment, fecal microbiota transplantation (FMT) is administered to restore healthy gut microbiota. FMT is delivered primarily via encapsulated microbiota capsules, with alternative routes including colonoscopy, gastroscopy, nasojejunal tube, or rectal enema if capsules are contraindicated. A second FMT dose is given 7 days after the first, either as daily capsules over six days or as a single endoscopic administration. This approach aims to reduce CDI recurrence by combining targeted antibiotic reduction of pathogens with microbiome restoration.
  Other Names: Vancomycin short-course pretreatment
  Arms: FECAL MICROBIOTA TRANSPLANTATION (with vancomycin short pretreatment phase)
Drug: Fidaxomicin — Participants receive a 10-day course of fidaxomicin administered orally at a dose of 200 mg twice daily. Fidaxomicin is a narrow-spectrum macrocyclic antibiotic specifically targeting Clostridioides difficile with minimal impact on the normal gut microbiota. This monotherapy aims to eradicate C. difficile infection while preserving the intestinal microbiome, thereby reducing the risk of recurrence. No additional interventions are provided during the treatment period. Biological samples are collected before and after treatment to evaluate clinical response, safety, and microbiome changes.
  Arms: ANTIBIOTICS ONLY - FIDAXOMICIN
Drug: Vancomycin (VAN) treatment — Participants receive a 10-day course of oral vancomycin at a dose of 125 mg four times daily. Vancomycin is a broad-spectrum glycopeptide antibiotic commonly used as standard-of-care therapy for Clostridioides difficile infection. This monotherapy aims to eradicate C. difficile by reducing bacterial load in the colon. No additional interventions are applied during the treatment period. Biological samples are collected before and after treatment to monitor clinical outcomes, safety, and changes in the gut microbiome.
  Arms: ANTIBIOTICS ONLY - VANCOMYCIN

SUMMARY:
The STOP-CDI study is a multicenter, randomized, open-label, three-arm clinical trial comparing the efficacy of fecal microbiota transplantation (FMT) preceded by vancomycin, fidaxomicin monotherapy, and standard-of-care vancomycin in preventing recurrence of Clostridioides difficile infection (CDI) in high-risk adult patients.

CDI is a common healthcare-associated infection with rising incidence and high recurrence rates, particularly in elderly and immunocompromised individuals. While current guidelines recommend fidaxomicin as first-line therapy, its availability and reimbursement remain limited in some healthcare systems. FMT, although effective, is not widely implemented as first-line treatment. This study addresses the need for comparative, real-world data to inform treatment decisions for patients at high risk of severe or recurrent CDI.

Eligible participants include adults aged ≥65 years or younger patients with specific risk factors such as multiple comorbidities, prior CDI episodes, recent hospitalization, use of non-CDI antibiotics, or PPI therapy. Participants will be randomized in a 2:1:1 ratio to one of three treatment arms: (1) vancomycin plus FMT, (2) fidaxomicin, or (3) vancomycin alone. FMT is administered via capsules or, if necessary, alternative endoscopic routes.

The primary endpoint is CDI recurrence within 12 weeks following the initial treatment. Secondary endpoints include clinical cure, safety, and global cure. Exploratory analyses will assess microbiome changes and potential genomic predictors of response. A total of 424 participants will be enrolled across 10 clinical sites in Poland.

The study aims to provide robust, comparative evidence to support clinical guidelines and improve outcomes for patients with CDI, particularly in healthcare systems with limited access to novel therapies.

DETAILED DESCRIPTION:
Clostridioides difficile infection (CDI) represents a persistent and growing challenge in modern healthcare, particularly among elderly, hospitalized, and immunocompromised patients. Despite the existence of evidence-based therapeutic guidelines, recurrence rates remain unacceptably high, often leading to cycles of reinfection and retreatment. These recurrent episodes are associated with increased morbidity, reduced quality of life, higher healthcare costs, and, in some cases, life-threatening complications.

While therapies such as fidaxomicin and fecal microbiota transplantation (FMT) have demonstrated superior efficacy in reducing recurrence compared to traditional vancomycin, access to these interventions remains inconsistent. Fidaxomicin is often restricted due to its high cost and limited reimbursement, while FMT-though highly effective-is not yet widely integrated into early-line treatment pathways, largely due to regulatory and logistical barriers, including donor screening, manufacturing infrastructure, and clinician training.

The STOP-CDI study is a multicenter, randomized, open-label, three-arm research experiment designed to directly compare the effectiveness of three therapeutic strategies in preventing recurrent CDI (rCDI) in a real-world, high-risk adult population. The project addresses key gaps identified by international societies such as ESCMID, which emphasize the need for high-quality, head-to-head comparative research in CDI management.

The primary objective is to determine which of the following approaches most effectively prevents CDI recurrence within 12 weeks after treatment completion:

1. Short-course oral vancomycin followed by FMT
2. Fidaxomicin monotherapy
3. Standard-of-care oral vancomycin

Participants will be randomized in a 2:1:1 allocation ratio, favoring the vancomycin plus FMT group to enable robust analysis of this relatively underutilized intervention. FMT is administered either as oral capsules containing freeze-dried donor microbiota or, when oral intake is not possible, through endoscopic routes such as colonoscopy or nasoenteric tubes. All FMT materials are sourced from rigorously screened donors under standardized laboratory protocols.

The study population includes 424 adult participants across 10 clinical sites in Poland, with recruitment targeting:

Adults aged 65 years or older, or

Younger adults with clearly defined risk factors for severe or recurrent CDI, such as:

* Multiple comorbidities (e.g., diabetes, malignancy, chronic kidney disease),
* Prior CDI episodes,
* Recent hospitalization,
* Use of non-CDI antibiotics,
* Ongoing proton pump inhibitor (PPI) therapy,
* Immunosuppressive treatment.

The primary endpoint of the experiment is CDI recurrence within 12 weeks following treatment, defined by return of symptoms (e.g., diarrhea) and laboratory confirmation of C. difficile toxin. Secondary endpoints include:

1. Initial clinical cure (symptom resolution at the end of therapy),
2. Global cure (clinical cure without recurrence),
3. Time to recurrence,
4. Safety and adverse event reporting,
5. Patient-reported outcomes, including quality-of-life metrics,
6. Healthcare resource utilization and cost-related measures.

In addition to clinical outcomes, the study includes a comprehensive biosample collection strategy for mechanistic and exploratory analyses. Longitudinal sampling of stool, blood, urine, and saliva will allow for in-depth evaluation of:

* Microbiome composition and dynamics,
* Inflammatory and immunological markers,
* Metabolomic profiling,
* Host genetic and genomic predictors of response or recurrence.

These exploratory analyses are intended to improve understanding of host-microbiota interactions in CDI and identify potential biomarkers for personalized treatment approaches.

The sample size of 424 has been statistically powered to detect an absolute difference of at least 15 percentage points in recurrence rates between the FMT group and standard vancomycin, with 80% power and a two-sided significance level of 0.05. This allows for subgroup analyses stratified by age, comorbidities, severity of CDI, and baseline risk factors.

Although the study is open-label, outcome assessment procedures include blinded adjudication by an independent clinical review board to minimize bias. In addition, centralized data monitoring and periodic safety reviews will be conducted to ensure compliance with ethical standards and protocol fidelity.

The STOP-CDI experiment is designed not only to assess comparative efficacy but also to explore real-world feasibility, implementation barriers, and economic considerations associated with newer CDI treatments. It aims to provide decision-makers and clinicians with relevant, actionable evidence that reflects the constraints and opportunities present in everyday clinical practice-particularly in healthcare systems with limited access to novel therapies like fidaxomicin or bezlotoxumab.

Ultimately, the results of this research are expected to guide more personalized, effective, and practical strategies for managing CDI, reducing the burden of recurrence, and improving patient outcomes in diverse clinical and economic contexts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years or older OR individuals aged 18 to 64 years who meet at least one of the following criteria:
* Presence of at least two comorbid chronic diseases from the groups of cardiovascular diseases, respiratory system diseases, gastrointestinal diseases, autoimmune diseases, cancers, chronic kidney and genitourinary diseases, immunodeficiencies, diabetes, and metabolic diseases,
* Previous episodes of CDI,
* Healthcare-associated CDI and/or hospitalization within the last three months,
* Concurrent use of antibiotics other than CDI treatment after CDI diagnosis,
* Use of proton pump inhibitors (PPIs) started during or after CDI diagnosis.
* Documented Clostridioides difficile infection, defined according to ESCMID as:

Diagnosis of diarrhea associated with C. difficile defined by:

* > 3 unformed stools (or >200 ml of unformed stool in patients with stool collection devices) within 24 hours before randomization AND
* Clinical signs consistent with CDI and microbiological evidence of free C. difficile toxins in an enzyme immunoassay (EIA) without justified evidence of another cause of diarrhea OR
* Clinical picture consistent with CDI and positive nucleic acid amplification test (NAAT; PCR) preferably with low cycle threshold (Ct) value, or positive toxigenic C. difficile culture OR
* Pseudomembranous colitis diagnosed during endoscopy or colectomy combined with a positive test for toxigenic C. difficile.
* No more than 24 hours of prior treatment with vancomycin, metronidazole, or fidaxomicin.
* Absolute neutrophil count in peripheral blood within 3 days before intervention > 500/µl.
* Ability to swallow large capsules (using test capsules) or no contraindications for FMT via nasojejunal tube, gastroscopy, colonoscopy, or rectal enema.
* Provided informed consent for participation in the clinical study.

Exclusion Criteria:

* Lack of consent to participate in the study or absence of logical contact without possibility of obtaining consent from an authorized person,
* More than 24 hours of prior treatment with vancomycin, metronidazole, or fidaxomicin,
* On the day of inclusion (up to 3 days before starting intervention) absolute neutrophil count in blood <500 cells/µl or expected drop to this level within the next 2 days,
* Diagnosed HIV infection with CD4 lymphocyte count <250 cells/µl,
* Inability to swallow large capsules (failed test capsule use) or contraindications for FMT via upper or lower gastrointestinal tract, including gastrointestinal perforation, anal atresia, discontinuity of the gastrointestinal tract, and others,
* Known presence of other pathogens in stool known to cause diarrhea,
* Life expectancy <3 months,
* Life-threatening CDI (fulminant at diagnosis - especially with septic shock),
* Total or subtotal colectomy, ileostomy, or colostomy,
* Unwillingness or inability to comply with protocol requirements, including any condition (physical, mental, or social) that may affect the participant's ability to adhere to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of Clostridioides difficile infection (CDI) within 12 weeks after treatment | 12 weeks (90 days) after treatment completion
  Proportion of patients experiencing a new episode of CDI, defined as recurrent diarrhea with confirmed C. difficile infection, within 12 weeks (90 days) after initial clinical cure following intervention.

SECONDARY OUTCOMES:
Initial Clinical Cure Rate | Up to 10 days from treatment initiation
  Proportion of patients achieving initial clinical cure, defined as resolution of diarrhea for at least 2 consecutive days during or after completion of standard antibiotic therapy.
Sustained clinical cure rate at 8 weeks post-treatment | 8 weeks (60 days) after treatment completion
  Percentage of patients with no recurrence of CDI symptoms and sustained clinical cure (no diarrhea) within 8 weeks (60 days) after completing therapy, confirmed by patient diary and clinical evaluation.
Recurrent CDI Rate at 8 Weeks | 8 weeks (60 days) after completion of therapy
  Proportion of patients experiencing a recurrence of Clostridioides difficile infection (CDI), defined as a new episode of diarrhea caused by C. difficile within 8 weeks (60 days) after initial clinical cure, confirmed by patient diary and clinical evaluation.
Sustained Clinical Cure Rate (Complete Cure) | 8 weeks (60 days) after treatment completion
  Proportion of patients with initial clinical cure and no recurrence of CDI symptoms for 8 weeks (60 days) after completing therapy.
Sustained Clinical Cure Rate (Durable Cure) | 12 weeks (90 days) after treatment completion
  Proportion of patients with initial clinical cure and no recurrence of CDI for 12 weeks (90 days) after completing therapy.
Rate of Treatment-Resistant CDI | Up to 10 days from treatment initia
  Proportion of patients with refractory CDI, defined as persistent diarrhea despite standard antibiotic therapy (vancomycin or fidaxomicin).
Incidence of Adverse Events | Up to 90 days after treatment
  Proportion of patients experiencing adverse events during the course of treatment and follow-up period. Safety will be assessed based on clinical examination and laboratory findings.

OTHER OUTCOMES:
Changes in gut microbiota diversity and composition after FMT | Baseline, Day 7, Day 14, and Weeks 4, 8, and 12 post-treatment
  Assessment of the diversity and composition of the intestinal microbiota before and after fecal microbiota transplantation using metagenomic sequencing, to evaluate microbiota restoration.

IPD SHARING:
Plan to Share IPD: Yes
Yes, individual participant data (IPD) will be shared with other researchers. Data sharing will be conducted only after the signing of a confidentiality agreement (non-disclosure agreement) to ensure the privacy and protection of participant information. Access to the data will be granted upon reasonable request and subject to approval by the study sponsor and ethics committee.